CLINICAL TRIAL: NCT05753527
Title: The Effect of Progressive Relaxation Exercises Applied Before Simulation Training on State Anxiety, Student Satisfaction and Perceived Stress Level of Nursing Students
Brief Title: The Effect of Progressive Relaxation Exercises on Anxiety, Satisfaction and Stress Levels Before Simulation Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nuh Naci Yazgan University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, DİDEM KAYA, Assistant Professor Doctor, Nuh Naci Yazgan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NuhNaciYazganUdkaya01
Record Dates: First submitted 2023-01-23; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Anxiety; Stress; Satisfaction; Relaxation; Joint, Congenital; Simulation
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive relaxation exercise group (Experimental): The students in the intervention group will be given progressive relaxation exercises before the simulation application. Before and after the simulation, vital signs will be taken and scales will be applied.
  Interventions: Behavioral: Progressive Relaxation Exercises
- The group not applied progressive relaxation exercise (No Intervention): The students in the control group will be taken into the simulation application without applying relaxation exercises. Before and after the simulation application, vital signs will be taken and scales will be applied.

INTERVENTIONS:
Behavioral: Progressive Relaxation Exercises — Deep abdominal breathing will be done three times and the breath will be given slowly. The fists will be clenched, keep the fists clenched in this way for 7-10 seconds, and then release them for 15-20 seconds. By opening the arms to the side and locking the elbows, the triceps muscle will be stretched and relaxed. The forehead muscles by raising the eyebrows The eyes will be closed and relaxed. The mouth will be opened and closed. The head will be stretched back and relaxed. The shoulders will be lifted and relaxed. Both hips will be tightened and relaxed by bringing them closer together. The thigh muscles will be tightened and relaxed.
  Arms: Progressive relaxation exercise group

SUMMARY:
The simulation-based learning method causes a sense of anxiety in students. Studies have shown that progressive relaxation exercises have a positive effect on anxiety. This study, will be tried to determine the effect of the progressive relaxation exercises applied to the students before the simulation training on anxiety, student satisfaction, and stress.

This study is an intervention study with a pretest-posttest control group. Before the study, Personal Information Form, State Anxiety Scale, Student Satisfaction and Self-Confidence in Learning Scale, Perceived Stress Scale for Nursing Students, and Students' Vital Findings Evaluation Form will be applied. After applying progressive relaxation exercises to the intervention group, they will be taken to the simulation laboratory. The control group will be taken to the simulation laboratory without any intervention. After the simulation application, the scales will be re-applied and the vital signs of the students will be measured again.

DETAILED DESCRIPTION:
Location of the research: The research was planned to be conducted at Hacettepe University Faculty of Nursing. There is a simulation laboratory in the department to enable students to perform their professional skills in a high-reality environment. In the laboratory, there are all kinds of equipment that a clinic should have, such as a medium reality simulation manikin, nurse's desk, patient bed, monitor, bedside oxygen systems, treatment, and emergency car. Lab; It consists of 3 parts application room, control room, and analysis room.Time of the research: The research will start after the approval of the ethics committee and institutional permissions. The implementation phase of the research is planned to be completed within 3 months. The universe of the research, the sample, the research group: The universe of the research; will consist of students studying in the 2nd year of the Faculty of Nursing. The main purpose of choosing this student group is that it is a group of students who have successfully completed the applied basic courses such as Internal Medicine Nursing and Surgical Nursing in the 2nd year, have basic knowledge and skills on illness and nursing care, but still do not have sufficient equipment in terms of intervening with the patient. In this student group, it was thought that when they were at the beginning of education and practices, progressive relaxation exercises application in reducing the anxiety they experienced during simulation training and increasing their learning satisfaction, raising awareness in this field and the use of this method in the further education processes would make significant contributions to student education. In this study, with the aim of determining the minimum sample size, the sample size was determined by considering the optimum sample numbers as a result of examining the sample sizes in which data saturation was reached in similar studies in the literature. According to this, after the power analysis, it was determined that a total of 27 people in each group should be required for multiple variance analysis in repeated measurements in a 2x2 factorial pattern between groups, with 80% power and a 5% margin of error. In the research, students who applied progressive relaxation exercises and simulation applications together will form the intervention group, and students who only participated in the simulation application will form the control group.

Type of the study: The research was planned in a randomized controlled design with the aim of determining the effect of progressive relaxation exercises applied before the simulation training on the state anxiety, student satisfaction, and perceived stress level of nursing students.

Application of Research An acquaintance and information meeting will be held before the progressive relaxation exercises sessions for students who meet the research criteria and agree to participate in the study. At the meeting, students will also be informed about the research and progressive relaxation exercises and their written informed consent will be obtained.

The data will be collected through the face-to-face interview technique, the application of progressive relaxation exercises, the data collection form, and scales developed by the researchers. The evaluations of the students in terms of physical parameters (vital signs) will be measured by the same researcher as pulse, respiratory rate, and blood pressure, respectively. Measurements will be taken repeatedly, before and after the simulation application, and the obtained values will be recorded. Students will be assigned to groups by simple random randomization method. In order to prevent the dependency relationship between students and researchers and to provide blinding between researchers, information about participation in the research will be made by the researcher who will carry out the progressive relaxation exercises application, and it will be especially emphasized that the student's acceptance or refusal to participate in the research will not affect their success grades. In this way, researchers other than the researcher who will apply the progressive relaxation exercises will continue the simulation training routinely without knowing which group the students are in. The days and time intervals of progressive relaxation exercise sessions will be determined with the students who will be in the intervention group in the research.

Pre-Test Before the simulation application and progressive relaxation exercises sessions, the State Anxiety Scale and the Perceived Stress Scale for Nursing Students will be administered to the students in both groups and their vital signs will be measured.

Intervention for the Intervention Group After the pre-test, progressive relaxation exercises will be applied to the students in the progressive relaxation exercises+simulation application group in an appropriate area in the Faculty of Nursing, and then the students will be taken to the simulation laboratory to perform the simulation application. An evaluation/analysis session will then be held.

Things to Do for the Control Group After the pre-test, the students in the control group will be given a simulation application in the simulation laboratory of the Faculty of Nursing by the researcher in the research team. An evaluation/analysis session will then be held.

Within the scope of the simulation application; The ideal number of students to take part in each simulation was determined to be 5. 2 days before the simulation day, all students will be given the necessary materials to prepare for the simulation application. On the day of the simulation, the researchers responsible for the simulation application will introduce the environment and the tools and equipment they will use in the simulation application in order for the students to make preliminary preparations. It will take a total of 60 minutes, including preliminary information (10 minutes), simulation time (15 minutes), and evaluation/analysis session (35 minutes).

Final Test After the progressive relaxation exercises and simulation application are completed by the researchers, the State Anxiety Scale, Student Satisfaction and Self-Confidence Scale in Learning, and Perceived Stress Scale for Nursing Students will be re-applied to the students and vital signs will be re-measured and recorded.

Analysis of the data:

The data to be obtained from the research will be evaluated by transferring them to the Statistical Packages for the Social Sciences Statistics 25 program. While evaluating the study data, descriptive statistics (mean, standard deviation, median, minimum, maximum) for continuous variables and frequency distribution for categorical variables will be given. The Mann-Whitney U Test will be used for the difference between two independent groups, and the Pearson correlation test will be used for the relationship between the scale scores. The significance level will be taken as p<0.05.

In addition to these evaluations; Per Protocol Analysis (PP) and Intention to Treat (ITT) analysis will also be performed. Per protocol, analysis is a method in which only the intervention groups are included in the analysis in intervention studies. Per protocol, the analysis reflects actual response performance. However, in cases where the losses are not random, there is a significant risk of bias. Therefore, the combined use of PP analysis and ITT is a recommended method to check the reliability of the results. ITT is a basic method used to maintain randomization and avoid bias on dropout. The ITT analysis revealed separation, non-compliance, whether or not to receive the treatment/intervention, etc. after randomization. It is defined as the inclusion of each participant in the analysis in the group to which they are assigned, without considering any justification. Researchers need to use at least one of the many statistical strategies to complete missing data (30). In addition, repeated assessments (State Anxiety Scale, Student Satisfaction and Self-Confidence in Learning Scale, and Perceived Stress Scale for Nursing Students) made in the research will be made by two researchers, and the fit (fisher's kappa) statistic will be used to evaluate the agreement.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer students aged 18 and over will be included in the study.

Exclusion Criteria:

* Using any medication that affects the heart rate,
* Having any psychiatric disease such as anxiety disorder,
* Students who do not accept to participate in the research will not be included in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Scale | It will be applied to the students just before simulation and after completing the training on the same day (each session is 60 minutes). Change from baseline State Anxiety Scale scores at the end of 60 minutes.
  It is an inventory developed to measure state and trait anxiety. Inventory is used to determine how an individual feels at a particular moment and in a situation. The scale is a very sensitive measurement tool for evaluating abruptly changing emotional reactions. The lowest total score that can be obtained from the State Anxiety Scale is 20, and the highest total score is 80. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety. The final result is the individual's state anxiety score. The scale is a very sensitive measurement tool for evaluating abruptly changing emotional reactions.
Student Satisfaction and Self-Confidence in Learning Scale | It will be applied to the students just before simulation and after completing the training on the same day (each session is 60 minutes). Change from baseline Student Satisfaction and Self-Confidence in Learning Scale scores at the end of 60 minutes.
  This scale, which is widely used to evaluate students' attitudes and beliefs about simulation, was published by the National League for Nurses. The highest total score that can be obtained from the scale is 65, and the lowest is 13. The high score that can be obtained from the total of the scale indicates high satisfaction and self-confidence.
Perceived Stress Scale for Nursing Students | It will be applied to the students just before simulation and after completing the training on the same day (each session is 60 minutes). Change from baseline Perceived Stress scores at the end of 60 minutes.
  The scale aims to measure the level of stress perceived by the students. The scale has six sub-dimensions (Stress caused by lack of professional knowledge and skills, Stress experienced while caring for the patient, Stress caused by homework and workload, Stress caused by instructors and nurses, Stress caused by the environment, Stress caused by peers and daily life). The total score of the scale ranges from 0 to 116. A high score indicates a high level of stress.
Change from Baseline Pulse Rates at 60 minutes | The pulse will be measured just before simulation training and after completing the training on the same day (each session is 60 minutes). Change from baseline pulse rates at the end of 60 minutes.
  The pulse rates of all students will be measured and recorded just before simulation training and after completing the training on the same day (each session is 60 minutes)
Change from Baseline Blood Pressure at 60 minutes | The blood pressure will be measured just before simulation training and after completing the training on the same day (each session is 60 minutes). Change from baseline blood pressure values at the end of 60 minutes.
  The blood pressure of all students will be measured and recorded just before simulation training and after completing the training on the same day (each session is 60 minutes)
Change from Baseline Respiratory Rates at 60 minutes | The respiratory rate will be measured just before simulation training and after completing the training on the same day (each session is 60 minutes). Change from baseline respiratory rate values at the end of 60 minutes.
  The respiratory rates of all students will be measured and recorded just before simulation training and after completing the training on the same day (each session is 60 minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Didem Kaya, Kocasi̇nan, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study results will be shared with other researchers.

REFERENCES:
- [Background] Abraham, C. M., & de Cordova, P. B. (2019). Simulation Activity and Inter-Professional Education in Pre-Licensure Nursing Programs in New Jersey: A 3 Year Trend Analysis. Teaching and Learning in Nursing, 14(3), 166-172.
- [Background] Jeffries, P. (2007). Simulation in Nursing Education: From Conceptualization to Evaluation. New York, NY: National League for Nursing.
- [Background] Mıdık, Ö., Kartal, M. (2010). Simülasyona dayalı tıp eğitimi. Marmara Medical Journal. 23(3): 389-99.
- [Background] Groom, A.J., Henderson, D., Sittner, J.B. (2013). National league for nursing jeffries simulation framework state of the science project:simulation design characteristics., Clinical Simulation in Nursing, 10(7): 337-344.
- [Background] Lewis R, Strachan A, Smith MM. Is high fidelity simulation the most effective method for the development of non-technical skills in nursing? A review of the current evidence. Open Nurs J. 2012;6:82-9. doi: 10.2174/1874434601206010082. Epub 2012 Jul 27. PMID 22893783
- [Background] Gosselin, K. P., Holland, B., Mulcahy, A., Williamson, S., & Widacki, A. (2016). Music for anxiety reduction and performance enhancement in nursing simulation. Clinical Simulation in Nursing, 12(1), 16-23.
- [Background] Nielsen, B., & Harder, N. (2013). Causes of student anxiety during simulation: What the literature says. Clinical Simulation in Nursing, 9(11), e507-e512.
- [Background] Yockey, J., & Henry, M. (2019). Simulation Anxiety across the Curriculum. Clinical Simulation in Nursing, 29, 29-37.
- [Background] Beischel KP. Variables affecting learning in a simulation experience: a mixed methods study. West J Nurs Res. 2013 Feb;35(2):226-47. doi: 10.1177/0193945911408444. Epub 2011 May 18. PMID 21593285
- [Background] Horsley, T. L., & Wambach, K. (2015). Effect of nursing faculty presence on students' anxiety, self-confidence, and clinical performance during a clinical simulation experience. Clinical Simulation in Nursing, 11, 4-10.
- [Background] Lai HL, Chen PW, Chen CJ, Chang HK, Peng TC, Chang FM. Randomized crossover trial studying the effect of music on examination anxiety. Nurse Educ Today. 2008 Nov;28(8):909-16. doi: 10.1016/j.nedt.2008.05.011. Epub 2008 Jul 1. PMID 18597899
- [Background] Horsley, T. L., & Wambach, K. (2015). Effect of nursing faculty presence on students' anxiety, self-confidence, and clinical performance during a clinical simulation experience. Clinical Simulation in Nursing, 11(1), 4-10.
- [Background] Moscaritolo LM. Interventional strategies to decrease nursing student anxiety in the clinical learning environment. J Nurs Educ. 2009 Jan;48(1):17-23. doi: 10.3928/01484834-20090101-08. PMID 19227751
- [Background] Martha L. Carver BSN, Maureen O'Malley PhD, Progressive muscle relaxation to decrease anxiety in clinical simulations, Teaching and Learning in Nursing, 2015, 10:57-62.
- [Background] Torabizadeh C, Bostani S, Yektatalab S. Comparison between the effects of muscle relaxation and support groups on the anxiety of nursing students: A randomized controlled trial. Complement Ther Clin Pract. 2016 Nov;25:106-113. doi: 10.1016/j.ctcp.2016.09.001. Epub 2016 Sep 7. PMID 27863599
- [Background] Dehghan-Nayeri N, Adib-Hajbaghery M. Effects of progressive relaxation on anxiety and quality of life in female students: a non-randomized controlled trial. Complement Ther Med. 2011 Aug;19(4):194-200. doi: 10.1016/j.ctim.2011.06.002. Epub 2011 Jul 12. PMID 21827933
- [Background] Spielberger CD, Gorsuch RL, Lushene RE, 1970. STAI. Manual for the State-Trait Anxiety Inventory (Self Evaluation Questionnaire). Palo Alto California: Consulting Psychologist, 22, 1-24.